CLINICAL TRIAL: NCT06912399
Title: Effect of Transauricular Vagus Nerve Stimulation on Postoperative Pain Management in Video Assisted Thoracic Surgery: a Randomized Controlled Clinical Trial
Brief Title: Effect of Transauricular Vagus Nerve Stimulation on Postoperative Pain Management in Video Assisted Thoracic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K7040
Record Dates: First submitted 2025-03-19; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain, Acute; VATS
Keywords: TaVNS; Postopearvie pain; VATS
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- taVNS group. (Experimental): Paticipants in this arm will undergo a 2-hour intervention of taVNS on the first postoperative day.
  Interventions: Device: Transauricular Vagus Nerve Stimulation
- sham-taVNS group. (Sham Comparator): Paticipants in this arm will undergo a 2-hour sham-intervention of taVNS on the first postoperative day.
  Interventions: Device: Sham Transauricular Vagus Nerve stimulation

INTERVENTIONS:
Device: Transauricular Vagus Nerve Stimulation — Participants enrolled will have a commercial transcutaneous electrical nerve stimulation unit (tVNS501,RISHENA,Changzhou,China) attached to their left outer ear after VATS. The stimulation pulses will target at the cymba concha which is 100% dominated by the auricular branch of the vagus nerve. Stimulation pulses will be 25Hz in frequency according to current clinical research, 500µs in pulse width which has been suggested to be most biologically active, with its amplitude increasing to the maximum amount that the patients can tolerate without pain.
  Other Names: taVNS
  Arms: taVNS group.
Device: Sham Transauricular Vagus Nerve stimulation — The only thing differs with the taVNS group is that the device will automatically shut down after running for 15 seconds.
  Other Names: Sham-taVNS
  Arms: sham-taVNS group.

SUMMARY:
Transcutaneous auricular vagus nerve stimulation (taVNS) is a novel pain management technique that has gained popularity in recent years due to its non-invasive nature and ease of operation. Current literature has substantiated its efficacy in managing pain syndromes and chronic pain. However, there is a paucity of evidence regarding its effectiveness in treating acute postoperative pain. This project aims to explore the efficacy of taVNS in postoperative pain management, with a focus on video-assisted thoracic surgery(VATS). The investigators have designed a double-blind, single-center, randomized controlled clinical trial, planning to enroll 116 patients scheduled to undergo VATS(including segmentectomy or lobectomy) under general anesthesia at Peking Union Medical College Hospital. Participants will be divided into an intervention group (receiving taVNS) and a sham intervention group (receiving sham-taVNS), and will undergo a 2-hour intervention on the first postoperative day. The primary outcome is the pain relief rate, defined as a reduction of 15mm or 30% in the VAS (1-100mm) score immediately before and after the intervention on the first postoperative day. Secondary outcomes include: the proportion of patients with inadequate analgesia within three days after intervention; the difference in VAS scores immediately before and after the intervention on the first postoperative day; the incidence of opioid-related and taVNS-related side effects from the first to the third postoperative day after intervention; the number of effective and ineffective PCA presses (if used) from the first to the third postoperative day after intervention; the specifics and frequency of additional analgesic measures taken by patients from the first to the third postoperative day after intervention; the difference in RCSQ scores on the night of surgery and the night after intervention; and the probability of patients experiencing surgery-related pain three months after surgery. Follow-up period for this study will be three months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. ASA classification I-III;
3. No prior taVNS treatment;
4. Scheduled to undergo VATS (including segmentectomy and lobectomy);
5. VAS ≥ 30 mm at any time on the day of surgery;
6. Patients and their families can understand the study design and are willing to cooperate and participate in the study.

Exclusion Criteria:

1. Psychiatric disorders or other conditions that prevent cooperation;
2. Long-term use of steroids or opioids;
3. Scheduled for bilateral VATS surgery;
4. History of thoracic surgery;
5. History of chronic pain, autoimmune diseases, or persistent infections.

Withdrawl Criteria:

1. Patient request;
2. Surgery cancellation or change in surgical method resulting in failure to meet inclusion criteria;
3. Severe perioperative complications and adverse events;
4. Severe intervention-related adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain Relief Rate | First postoperative day
  Pain relief rate is defined as a reduction of 15mm or 30% in the VAS (Visual Analogue Scale, 1-100mm) score immediately before and after the intervention on the first postoperative day

SECONDARY OUTCOMES:
The proportion of patients with inadequate analgesia within three days after intervention | Within three days after the intervention
  "Inadequate analgesia" is defined as: 1) VAS ≥ 40 mm at any time within three days after the intervention; or 2) the need for additional analgesic medication in the ward after the intervention, or the occurrence of ineffective PCA presses. Meeting either of the above criteria satisfies the definition.
The difference in VAS scores immediately before and after the intervention on the first postoperative day | First postoperative day
The incidence of opioid-related and taVNS-related side effects from the first to the third postoperative day after intervention | First to the third postoperative day
The number of effective and ineffective PCA attempts (if used) from the first to the third postoperative day after intervention | First to the third postoperative day
The specifics and frequency of additional analgesic measures taken by patients from the first to the third postoperative day after intervention | First to the third postoperative day
  The investigators will document any additional analgesic measures taken by the patients within three days after the intervention, including:
  The name, dosage, and administration method of analgesic medications; The formulation and settings of patient-controlled analgesia (PCA) pumps, along with the counts of effective and ineffective PCA attempts; Any physical analgesic measures employed.
The difference in RCSQ scores on the night of surgery and the night after intervention | First to second postoperative day
The probability of patients experiencing surgery-related pain three months after surgery | Three months after surgery
  The investigators will conduct a telephone follow-up with participants three months later to assess whether they still experience surgery-related pain after discharge. The outcome will be recorded as "yes" or "no" based on the patient's subjective description.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Considering patients' privacy and the measures for protecting participants, we do not plan to disclose patients' personal data.

REFERENCES:
- [Background] Gerner P. Postthoracotomy pain management problems. Anesthesiol Clin. 2008 Jun;26(2):355-67, vii. doi: 10.1016/j.anclin.2008.01.007. PMID 18456219
- [Background] Zhou Q, Yu L, Yin C, Zhang Q, Tai Y, Zhu L, Dong J, Wang Q. Effect of Transauricular Vagus Nerve Stimulation on Rebound Pain After Ropivacaine Single Injection Femoral Nerve Block for Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial. J Pain Res. 2022 Jul 14;15:1949-1958. doi: 10.2147/JPR.S370589. eCollection 2022. PMID 35860416
- [Background] Ayoo K, Mikhaeil J, Huang A, Wasowicz M. The opioid crisis in North America: facts and future lessons for Europe. Anaesthesiol Intensive Ther. 2020;52(2):139-147. doi: 10.5114/ait.2020.94756. PMID 32419434
- [Background] Costa V, Gianlorenco AC, Andrade MF, Camargo L, Menacho M, Arias Avila M, Pacheco-Barrios K, Choi H, Song JJ, Fregni F. Transcutaneous vagus nerve stimulation effects on chronic pain: systematic review and meta-analysis. Pain Rep. 2024 Aug 7;9(5):e1171. doi: 10.1097/PR9.0000000000001171. eCollection 2024 Oct. PMID 39131814
- [Background] Straube A, Eren O. tVNS in the management of headache and pain. Auton Neurosci. 2021 Dec;236:102875. doi: 10.1016/j.autneu.2021.102875. Epub 2021 Aug 31. PMID 34500261
- [Background] Pacheco-Barrios K, Gianlorenco AC, Camargo L, Andrade MF, Choi H, Song JJ, Fregni F. Transauricular Vagus Nerve Stimulation (taVNS) enhances Conditioned Pain Modulation (CPM) in healthy subjects: A randomized controlled trial. Brain Stimul. 2024 Mar-Apr;17(2):346-348. doi: 10.1016/j.brs.2024.03.006. Epub 2024 Mar 5. No abstract available. PMID 38453004
- [Background] Ramaswamy S, Wodehouse T. Conditioned pain modulation-A comprehensive review. Neurophysiol Clin. 2021 Jun;51(3):197-208. doi: 10.1016/j.neucli.2020.11.002. Epub 2020 Dec 14. PMID 33334645
- [Background] Kaniusas E, Kampusch S, Tittgemeyer M, Panetsos F, Gines RF, Papa M, Kiss A, Podesser B, Cassara AM, Tanghe E, Samoudi AM, Tarnaud T, Joseph W, Marozas V, Lukosevicius A, Istuk N, Sarolic A, Lechner S, Klonowski W, Varoneckas G, Szeles JC. Current Directions in the Auricular Vagus Nerve Stimulation I - A Physiological Perspective. Front Neurosci. 2019 Aug 9;13:854. doi: 10.3389/fnins.2019.00854. eCollection 2019. PMID 31447643
- [Background] Chen M, Yu L, Ouyang F, Liu Q, Wang Z, Wang S, Zhou L, Jiang H, Zhou S. The right side or left side of noninvasive transcutaneous vagus nerve stimulation: Based on conventional wisdom or scientific evidence? Int J Cardiol. 2015;187:44-5. doi: 10.1016/j.ijcard.2015.03.351. Epub 2015 Mar 23. No abstract available. PMID 25828310
- [Background] Wang Y, Li SY, Wang D, Wu MZ, He JK, Zhang JL, Zhao B, Hou LW, Wang JY, Wang L, Wang YF, Zhang Y, Zhang ZX, Rong PJ. Transcutaneous Auricular Vagus Nerve Stimulation: From Concept to Application. Neurosci Bull. 2021 Jun;37(6):853-862. doi: 10.1007/s12264-020-00619-y. Epub 2020 Dec 23. PMID 33355897
- [Background] Gentile F, Orlando G, Montuoro S, Ferrari Chen YF, Macefield V, Passino C, Giannoni A, Emdin M. Treating heart failure by targeting the vagus nerve. Heart Fail Rev. 2024 Nov;29(6):1201-1215. doi: 10.1007/s10741-024-10430-w. Epub 2024 Aug 9. PMID 39117958
- [Background] Ben-Menachem E, Revesz D, Simon BJ, Silberstein S. Surgically implanted and non-invasive vagus nerve stimulation: a review of efficacy, safety and tolerability. Eur J Neurol. 2015 Sep;22(9):1260-8. doi: 10.1111/ene.12629. Epub 2015 Jan 23. PMID 25614179
- [Background] Nicholson WC, Kempf MC, Moneyham L, Vance DE. The potential role of vagus-nerve stimulation in the treatment of HIV-associated depression: a review of literature. Neuropsychiatr Dis Treat. 2017 Jun 28;13:1677-1689. doi: 10.2147/NDT.S136065. eCollection 2017. PMID 28721049
- [Background] Bonaz B. Enteric neuropathy and the vagus nerve: Therapeutic implications. Neurogastroenterol Motil. 2025 Aug;37(8):e14842. doi: 10.1111/nmo.14842. Epub 2024 Jun 14. PMID 38873822